CLINICAL TRIAL: NCT00035269
Title: Linezolid in the Treatment of Penicillin-Resistant Streptococcus Pneumoniae Pneumonia: An Open-Label, Non-Comparator Study
Brief Title: New Antibiotic to Treat Patients With Community-acquired Pneumonia Due to a Specific Bacteria (S. Pneumoniae Pneumonia)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: M12600071; A5951056
Record Dates: First submitted 2002-05-02; First posted 2002-05-03 (Estimated); Last update posted 2011-04-26 (Estimated); Status verified 2011-04

CONDITIONS: Pneumonia, Pneumococcal; Community Acquired Infections; Gram-positive Bacterial Infections
Keywords: Pharmacia
MeSH Terms: conditions — Pneumonia, Pneumococcal; Community-Acquired Infections; Gram-Positive Bacterial Infections | interventions — Anti-Bacterial Agents

INTERVENTIONS:
Drug: Antibiotic

SUMMARY:
This study will treat patients who have a community-acquired pneumonia that is due to a specific bacteria (S. pneumoniae)

ELIGIBILITY:
Other specific inclusion/exclusion criteria may apply. In order to determine eligibility, further examination by the investigator is necessary.

Inclusion Criteria:

* Patients must have the signs and symptoms of pneumonia, with a chest xray showing a pneumonia.
* The patient must have S. pneumoniae (a specific bacteria) growing in sputum or blood to continue treatment.

Exclusion Criteria:

* Patients cannot have taken more than one day of another antibiotic before entering this study.
* Patients with HIV and a low CD4 count are excluded.

Min Age: 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 230 (Actual)
Dates: Start 2001-12; Study Completion 2003-05 (Actual)

PRIMARY OUTCOMES:
To assess the microbiologic efficacy of linezolid in the treatment of patients with pneumonia caused by penicillin-resistant Streptococcus pneumoniae (PRSP).
Additionally, microbiologic efficacy will be assessed in all pneumonia patients infected with S pneumoniae SP) and in those infected with penicillin-sensitive (PSSP) and penicillin-intermediate (PISP) S pneumoniae.

SECONDARY OUTCOMES:
To assess clinical efficacy and safety in pneumonia patients infected with S pneumoniae.

CONTACTS AND LOCATIONS:
Locations (40):
- United States (32):
  - Research Center, Los Angeles, California
  - Research Center, Jacksonville, Florida
  - Research Center, Naples, Florida
  - Research Center, Savannah, Georgia
  - Research Center, Springfield, Illinois
  - Research Center, Baton Rouge, Louisiana
  - Research Center, Baltimore, Maryland
  - Research Center, Ann Arbor, Michigan
  - Research Center, Royal Oak, Michigan
  - Research Center, Springfield, Missouri
  - Research Center, Hackensack, New Jersey
  - Research Center, Newark, New Jersey
  - Research Center, Somerville, New Jersey
  - Research Center, Staten Island, New York
  - Research Center, Stony Brook, New York
  - Research Center, Columbus, Ohio
  - Research Center, Zanesville, Ohio
  - Research Center, Fleetwood, Pennsylvania
  - Research Center, Hershey, Pennsylvania
  - Research Center, Ninety Six, South Carolina
  - Research Center, Spartanburg, South Carolina
  - Research Center, Harrogate, Tennessee
  - Research Center, Jackson, Tennessee
  - Research Center, Knoxville, Tennessee
  - Research Center, Memphis, Tennessee
  - Research Center, Nashville, Tennessee
  - Research Center, Dallas, Texas
  - Research Center, Houston, Texas
  - Research Center, Lubbock, Texas
  - Research Center, Charlottesville, Virginia
  - Research Center, Richmond, Virginia
  - Research Center, Seattle, Washington
- Research Center, Bratislava, Slovakia
- Spain (5):
  - Research Center, Barcelona, Barcelona
  - Research Center, Mataró, Barcelona
  - Research Center, Girona, Girona
  - Research Center, Madrid, Madrid
  - Research Center, Móstoles, Madrid
- Taiwan (2):
  - Research Center, Kaohsiung City
  - Research Center, Taoyuan District